CLINICAL TRIAL: NCT04131153
Title: Percutaneous Ultrasound-guided "Three-step" Radiofrequency Ablation for Giant Hepatic Hemangioma: a Safe, Feasible and Effective New Technology
Brief Title: Percutaneous Ultrasound-guided "Three-step" Radiofrequency Ablation for Giant Hepatic Hemangioma
Acronym: RFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, fengkai, Principal Investigator, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180407
Record Dates: First submitted 2019-10-11; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Hepatic Hemangioma
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radiofrequency ablation group (Other): Conventional radiofrequency ablation procedures
  Interventions: Procedure: radiofrequency ablation
- Three-step radiofrequency ablation group (Experimental): After destroying the main blood supply of the tumor, extracting the blood in the tumor, reducing the blood flow in the tumor and shrinking the tumor volume, the remaining tumor was then treated with radiofrequency ablation, namely the "three-step" radiofrequency ablation with "one block, two inhalation and three damages".
  Interventions: Procedure: "three-step" radiofrequency ablation

INTERVENTIONS:
Procedure: "three-step" radiofrequency ablation — After destroying the main blood supply of the tumor, extracting the blood in the tumor, reducing the blood flow in the tumor and shrinking the tumor volume, the remaining tumor was then treated with radiofrequency ablation, namely the "three-step" radiofrequency ablation with "one block, two inhalation and three damages".
  Arms: Three-step radiofrequency ablation group
Procedure: radiofrequency ablation — Conventional radiofrequency ablation
  Arms: Conventional radiofrequency ablation group

SUMMARY:
Hepatic hemangioma is the most common benign tumor of the liver.For huge liver hemangioma, however, it need to use the conventional radiofrequency ablation can increase one-time ablation volume of radiofrequency electrode or enhance ablation power and extend the melting time, not only bring patients suffering discomfort, but easy to damage the adjacent organs, causing serious complications such as hemorrhage, perforation of gastrointestinal tract,acute renal failure .Therefore, the investigators have developed a new, standardized radiofrequency ablation for giant hepatic hemangioma to shorten the duration of treatment, reduce surgical complications and improve the surgical success rate.

The purpose of this study was to evaluate the safety, feasibility and efficacy of the new radiofrequency ablation (" three-step "radiofrequency ablation) in the treatment of giant hepatic hemangioma.

DETAILED DESCRIPTION:
Hepatic hemangioma is the most common benign tumor of the liver, with an incidence of 0.4-20% in the general population.For small and asymptomatic patients with hepatic hemangioma, regular reexamination is necessary without medical intervention.However, patients with giant hepatic hemangioma(diameter ≥ 5cm) may have symptoms such as abdominal pain, indigestion, jaundice, or rapid increase in lesion volume, or even spontaneous rupture and hemorrhage, which require active treatment.Currently, surgical resection is the most effective method for the treatment of hepatic hemangioma, but the incidence and mortality of related complications have been reported as high as 27% and 3% respectively

.Other alternative therapies, such as transcatheter arterial embolization, radiotherapy and steroid therapy, have also been reported for the treatment of hepatic hemangioma, but the efficacy is not satisfactory .

Percutaneous ultrasound-guided radiofrequency ablation is a safe and minimally invasive treatment with reliable efficacy. In recent years, this technique has been successfully applied in the treatment of hepatic hemangioma with a diameter of < 5cm.For huge liver hemangioma, however, need to use the conventional radiofrequency ablation can increase one-time ablation volume of radiofrequency electrode or enhance ablation power and extend the melting time, not only bring patients suffering discomfort, but easy to damage the adjacent organs, causing serious complications such as hemorrhage, perforation of gastrointestinal tract, acute renal failure .Therefore, the investigators have developed a new,standardized radiofrequency ablation for giant hepatic hemangioma to shorten the duration of treatment, reduce surgical complications and improve the surgical success rate.

The purpose of this study was to evaluate the safety, feasibility and efficacy of the new radiofrequency ablation (" three-step "radiofrequency ablation) in the treatment of giant hepatic hemangioma.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of hepatic hemangioma (more than two imaging evidences: enhanced ultrasound or enhanced CT and MRI), single tumor, 5-15cm in diameter;
2. The Child-Pugh grade A/B;
3. The ICG15 20% or less;
4. The eCOG score was 0;
5. The patients was persistent hemangioma-related abdominal pain or discomfort, and it has clear exclusion of other gastrointestinal diseases causing upper abdominal pain by gastroscopy;
6. The patients refused to receive surgical treatment, but agreed to receive radiofrequency ablation;
7. There were no other related diseases affecting RFA treatment.

Exclusion Criteria:

1. Multiple hepatic hemangioma lesions or single lesion < 5cm;
2. Severe primary organ failure, such as liver, kidney, heart, lung or brain;
3. Severe bleeding tendency, platelet count < 50 ×10^9/L, or prothrombin time extension > 18s;
4. Previous treatment of hepatic hemangioma (TACE, steroids, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Duration of Radiofrequency ablation | 60 minute
  Duration of Radiofrequency ablation
Duration of hospitalization | 7 day
  Duration of hospitalization

IPD SHARING:
Plan to Share IPD: No